CLINICAL TRIAL: NCT01212120
Title: The Foot in Your Nose Study: Links Between Nasal Staphylococcus Aureus Colonies and Diabetic Foot Lesion Infections
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: PHRC-I/2009/JPL-02; 2009-A00849-48 (Other: Afssaps, RCB number)
Record Dates: First submitted 2010-09-29; First posted 2010-09-30 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Diabetic Foot; Staphylococcus Aureus
Keywords: Diabetic foot
MeSH Terms: conditions — Diabetic Foot; Staphylococcal Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The DNA samples correspond to the bacteria present in the nose and feet of diabetic patients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients: All patients
  Interventions: Biological: Genetic profiling of bacterial cultures

INTERVENTIONS:
Biological: Genetic profiling of bacterial cultures — Genetic profiling of bacterial cultures harvested from both the nose and foot lesions of patients

SUMMARY:
The presence of S aureus in the nasal passages of diabetic patients may be a risk factor for diabetic foot lesion infections. Our aim is to compare the genetic profiles of S aureus strains found in the noses and on the foot lesions of diabetic patients. The investigators are also studying the virulence of these strains, the prevalance of S aureus at either site, and whether or not the quantity of S aureus found in the nose affects the risk for infection in foot lesions. The investigators also use this study to test the sensitivity and specificity of the GeneXpert system.

ELIGIBILITY:
Inclusion Criteria:

* Type 1 or 2 diabetic patients
* Patients consulting or hospitalized in the Diabetology departments of one of the participating centers
* Grade 2-4 ulcer on the foot or ankle (both primo and recurrent events are acceptable)

Exclusion Criteria:

* Patient refuses to participate
* Pregnant, parturient or breastfeeding women
* Patient does not have diabetic foot or arteritic
* Diabetic ulcer is located elsewhere than the foot or ankle
* The ulcer is non-swabbable
* Patient does not have social-security coverage
* Patient is under any type of guardianship

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult type 1 or 2 diabetic patients with grade 2-4 foot or ankle ulcers (first event or recurrence)
Sampling Method: Non-Probability Sample
Enrollment: 278 (Actual)
Dates: Start 2010-09; Primary Completion 2012-03-19 (Actual); Study Completion 2012-03-19 (Actual)

PRIMARY OUTCOMES:
Presence/absence of the same S. aureus genetic profile in the nose and on the foot lesion. | 3 hours
  Presence/absence of the same S. aureus genetic profile in the nose and on the foot lesion. Genetic profiles do not change with time. This is a transversal, pinpoint measure.

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Lavigne, MD PhD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (4):
- France (4):
  - CHU de Nîmes - Hôpital Universitaire Carémeau, Nîmes, Gard
  - CHU de Nîmes - Hôpital Universitaire de Réadaptation du Grau du Roi, Le Grau-du-Roi
  - APHM - Hôpital Nord, Marseille
  - CHU de Montpellier - Hôpital Lapeyronie, Montpellier

REFERENCES:
- [Result] Dunyach-Remy C, Courtais-Coulon C, DeMattei C, Jourdan N, Schuldiner S, Sultan A, Carriere C, Alonso S, Sotto A, Lavigne JP. Link between nasal carriage of Staphylococcus aureus and infected diabetic foot ulcers. Diabetes Metab. 2017 Apr;43(2):167-171. doi: 10.1016/j.diabet.2016.09.003. Epub 2016 Oct 5. PMID 27720361